CLINICAL TRIAL: NCT00156988
Title: The Effect of Two Versus Ten Days Application of Flammacerium in Partial Thickness Burns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Dutch Burns Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WO/P04.103; WO/P04.103
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Burns
Keywords: burns; partial thickness; cerium flamazine; randomised clinical trial
MeSH Terms: conditions — Burns | interventions — cerous nitrate, sulfadiazine silver drug combination

INTERVENTIONS:
Drug: cerium nitrate-silver sulfadiazine (cerium-flamazine)

SUMMARY:
The objective of the proposed study is to assess whether the application of flammacerium for 2 days is as good as, or even better than, the application of flammacerium for 10 days regarding woundhealing in partial thickness burns.

DETAILED DESCRIPTION:
Cerium is suggested to halt the cytokine cascade ensuing burn injury by binding the 'burn toxin' and, when used in combination with silver-sulfadiazine, may enhance its antibacterial effect. Since 1984, the combination of cerium and silver sulfadiazine, flammacerium, has been used in our centre. Current practice is to treat acute, non-facial, burns with daily cleaning and (re-)application of flammacerium for a total of ten days. However, prolonged application of cerium is thought to be unnecessary - it is effective in the early stages after injury- and prolonged application of silver sulfadiazine has a negative effect on wound healing. The objective of the proposed study is therefore, to assess whether the application of flammacerium for 2 days is as good as, or even better than, the application of flammacerium for 10 days regarding woundhealing in partial thickness burns.

ELIGIBILITY:
Inclusion Criteria:

* patients having partial thickness burns with TBSA of < 10%

Exclusion Criteria:

* patients not seen within 24 hours postburn
* patients with only facial burns
* patients with electrical or chemical burns
* patients or their parents/caregivers with mental or cognitive deficits that may interfere with providing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-03; Study Completion 2005-12

PRIMARY OUTCOMES:
number of days required for wound healing, judged clinically and assessed as both number of days till 95% and 100% re-epithelialisation by planimetry at the time the decision regarding surgery is made (8-10 pb) and as wounds are considered healed

SECONDARY OUTCOMES:
Wound colonisation, assessed by swabs taken at 0 or 3 days pb, 7 days pb and subsequently every 7 days until wounds are healed or treated surgically, and on indication

CONTACTS AND LOCATIONS:
Overall Officials: Marianne K Nieuwenhuis, PhD, Principal Investigator — Association Dutch Burns Centres
Locations (1):
- Burns Centre, Martini Hospital, Groningen, Netherlands